CLINICAL TRIAL: NCT00604136
Title: Treatment of Metastatic Melanoma Patients With Tumor Infiltrating Lymphocytes and IL-2 Following a Regimen of Non-myeloablative Lymphocyte Depleting Chemotherapy
Brief Title: Treatment of Metastatic Melanoma With Tumor Infiltrating Lymphocytes and IL-2 Following Lympho-depleting Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Michal Lotem, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS269- HMO-CTIL
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; tumor infiltrating lymphocytes; interleukin-2
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: tumor infiltrating lymphocytes — Patients will have a melanoma metastasis resected and cultured in IL-2 in vitro. Tumor infiltrating lymphocytes from these cultures will be assessed for tumor reactivity and those with such activity will be further expanded and adoptively transferred. Patients will receive a non-myeloablative lymphocyte-depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day x2 days IV)and fludarabine (25 mg/mE2/day IV x5days). Following this regimen, patients will receive an intravenous adoptive transfer of at least 10E9 tumor-reactive lymphocytes followed by high dose IL-2 (720,000 IU/kg/dose IV every 8 hours for up to 15 doses).

SUMMARY:
Prior preclinical and clinical studies have shown that tumors from patients with advanced melanoma contain tumor-infiltrating lymphocytes (TIL) with anti-tumor reactivity. These TIL can be expanded in the laboratory to large numbers, and reinfused to the patient. Using a chemotherapy regimen that selectively kills lymphocytes, a single institution Phase II study of 35 patients showed a 51% objective response rate to TIL and interleukin-2 injection. In the present trial we would like to investigate whether we can achieve similar results in a Hadassah Phase II study, and to determine the feasibility of applying this approach to patients with advanced melanoma who currently have few treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have metastatic melanoma with a resectable metastatic lesion of sufficient size and be willing to undergo such a resection for experimental purposes. For HLA-A0201+ patients, lesions must be > 1.5 cm in diameter and for HLA-A0201- patients, lesions must be > 3 cm in diameter.
* Patients must be > 18 years of age and must have measurable metastatic melanoma (in addition to the resected lesion).
* Patients of both genders must be willing to practice birth control during treatment and for four months after receiving the preparative regimen.
* Clinical performance status of ECOG 0, 1.
* Absolute neutrophil count greater than 1000/mm3 without support of filgrastim.
* Platelet count greater than 100,000/mm3.
* Serum ALT/AST less than three times the upper limit of normal.
* Serum creatinine less than or equal to 1.6 mg/dl.
* Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.
* Patients must be able to understand and sign the Informed Consent document

Exclusion Criteria:

* Tumor/TIL Harvest Exclusion Criteria:

  * Less than 4 weeks has elapsed since any prior systemic therapy or less than six weeks since prior nitrosourea therapy
  * Women who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
  * Life expectancy of less than three months.
  * Patients who have received prior treatment with anti-CTLA-4 antibody will be excluded unless a post anti-CTLA-4 antibody treatment colonoscopy was normal with normal colonic biopsies.
  * Patients who require immediate active treatment for symptomatic CNS lesions will not be eligible until after treatment of their symptomatic lesions.
* Cell Infusion Exclusion Criteria:

  * Less than 4 weeks has elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, or less than six weeks since prior nitrosourea therapy. All patients' toxicities must have recovered to a grade 1 or less or as specified in the eligibility criteria. Patients may have undergone minor surgical procedures or focal palliative radiotherapy (to non-target lesions) within the past 4 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.
  * Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
  * Life expectancy of less than three months.
  * Requirement for systemic steroid therapy.
  * Hemoglobin less than 8g/dl unable to be corrected with transfusion.
  * Any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
  * Any form of primary or secondary immunodeficiency. Must have recovered immune competence after chemotherapy or radiation therapy as evidenced by normal ANC > 1000/mm3 and absence of opportunistic infections. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Seropositive for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
  * Patients with hepatitis B or hepatitis C will be excluded.
* The following patients will be excluded because of inability to receive high dose interleukin-2:

  * Patients will be excluded if they have a history of major EKG abnormalities, symptoms of cardiac ischemia or arrhythmias and have a LVEF < 45% on a cardiac stress test (stress thallium, stress MUGA, dobutamine, echocardiogram or other stress test)
  * Similarly, patients who are 50 years old or greater with an LVEF < 45% will be excluded
  * Patients who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction will be excluded if they have an abnormal pulmonary function test as evidenced by a FEV1 < 60% predicted.
  * Patients who have received prior treatment with anti-CTLA-4 antibody will be excluded unless a subsequent colonoscopy was normal with normal colonic biopsies (to rule out colitis).
  * Patients who require immediate treatment for symptomatic CNS lesions will not be eligible until after treatment of their symptomatic lesions and resolution of symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
To determine the response rate of this approach when administered in our hospital | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel